CLINICAL TRIAL: NCT04856423
Title: Ultra-sensitivity Quantitative Fecal Immunochemical Test Improve Diagnostic Accuracy in Detecting Colorectal Advanced Adenoma and Colorectal Cancer: a Multicenter, Prospective Study
Brief Title: Ultra-sensitivity Quantitative Fecal Immunochemical Test in Detecting Colorectal Advanced Adenoma and Colorectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Collaborators: Shanghai Tongji Hospital, Tongji University School of Medicine (Other); Tianjin Medical University General Hospital (Other); Binzhou Medical University (Other); Weihai Municipal Hospital (Other); People's Hospital of Lixia District of Jinan (Unknown)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Other Study IDs: 2020SDU-QILU-1026
Record Dates: First submitted 2021-04-19; First posted 2021-04-23 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Colorectal Neoplasm
Keywords: Colorectal Neoplasm; Occult Bleeding; Quantitative fecal immunochemical test; Colorectal Cancer; Adenoma
MeSH Terms: conditions — Colorectal Neoplasms; Adenoma | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Us-qFIT group: People in this group will detect fecal hemoglobin concentration by us-qFIT before colonoscopy.
  Interventions: Diagnostic Test: The us-qFIT and colonoscopy with pathological examination

INTERVENTIONS:
Diagnostic Test: The us-qFIT and colonoscopy with pathological examination — Detect fecal hemoglobin concentration by us-qFIT before colonoscopy, detect colon lesions using colonoscopy and pathological examination.

SUMMARY:
Early detecting and removing of colorectal advanced adenomas can reduce the incidence of colorectal cancer. Because of the less bleeding of advanced adenomas, sensitivities of the common used quantitative fecal immunochemical tests (qFITs) are unsatisfying. Ultra-sensitivity qFIT(us-qFIT) can determine extremely low fecal hemoglobin concentration compared with the common used qFIT. This study will prove the diagnostic accuracy of us-qFIT in detecting colorectal advanced adenomas.

DETAILED DESCRIPTION:
Early detection of CRC in a curable stage can reduce mortality but not morbidity. The majority of colorectal cancer is thought to arise from precancerous lesions through the adenoma-carcinoma pathway. Detecting and removing of colorectal advanced adenomas can reduce incidence of colorectal cancer. Although colonoscopy is currently considered the most effective method for detecting advanced adenomas, individuals may be reluctant to undergo colonoscopy due to the uncomfortable feeling and the relatively high cost. Conversely, stool tests are relatively cheap and more readily accepted. Fecal immunochemical test (FIT) is economic and easy to use in colorectal cancer screening. However, the common used qFIT is insufficiently sensitive to the minor hemorrhage of advanced adenomas, and the sensitivity is about only 27% to 47%. To improve the detection rate of colorectal advanced adenoma, Ultra-sensitivity quantitative fecal immunochemical test (us-qFIT) improves technology and can detect fecal hemoglobin in extremely low concentration quantificationally. The investigators design this research to prove the diagnostic accuracy of us-qFIT in detecting colorectal advanced adenoma.

ELIGIBILITY:
Inclusion Criteria:

* 50-75 years old people;
* People sign an "informed consent form"

Exclusion Criteria:

* People with history of colorectal surgery;
* People with history of colorectal cancer;
* People with history of other diseases that may produce fecal blood, such as inflammatory bowel disease, ischemic enteritis, vascular alformation of intestine, intestinal tuberculosis or Non-Hodgkin's lymphoma involving digestive tract;
* People with symptoms including visible rectal bleeding, hematuria, hemorrhoid bleeds, severe and acute diarrhea and watery stool;
* People are in pregnancy, lactation or menstrual phase;
* People with severe congestive heart failure or other sever disease cause cannot tolerate colonoscopy.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Continuous participants intending to undergo colonoscopy and meet the inclusion and exclusion criteria from the 5 hospitals were enrolled.
Sampling Method: Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2021-04-19 (Actual); Primary Completion 2023-04-19 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
The accuracy of us-qFIT to diagnose colorectal advanced adenoma. | 24 months
  The sensitivity, specificity, positive predictive value and negative predictive value.

SECONDARY OUTCOMES:
The accuracy of us-qFIT to diagnose colorectal cancer. | 24 months
  The sensitivity, specificity, positive predictive value and negative predictive value.
The accuracy of us-qFIT to diagnose high-risk adenoma. | 24 months
  The sensitivity, specificity, positive predictive value and negative predictive value.
Develop a predictive model of advanced colorectal neoplasms which includes the value of us-qFIT. | 24 months
  Develop a predictive model of CRC or advanced colorectal neoplasm which includes qFIT, age ,sex, CRC family history, diet and so on.

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, PhD, Study Chair — Qilu Hospital of Shandong University
Locations (6):
- China (6):
  - Binzhou Medical University Hospotal, Binzhou, Shandong
  - People's Hospital of Lixia District of Jinan, Jinan, Shandong
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Weihai Municipal Hospital, Weihai, Shandong
  - Shanghai Tongji Hospital, Tongji University School of Medicine, Shanghai, Shanghai Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality